CLINICAL TRIAL: NCT03394326
Title: Implementing a Dietary Energy Density Intervention in Preschool Children
Brief Title: Eat Healthy for Families
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Delaware (Other)
Responsible Party: Principal Investigator, Shannon Robson, Principal Investigator, University of Delaware
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 1097650
Record Dates: First submitted 2018-01-03; First posted 2018-01-09 (Actual); Last update posted 2022-05-18 (Actual); Status verified 2022-05

CONDITIONS: Obesity, Childhood; Energy Density; Diet Quality
MeSH Terms: conditions — Pediatric Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- LOW-ED (Experimental): In the LOW-ED condition each participant will consume at least 10 low-ED foods/day (ED ≤1.0 kcal/g) and no more than 2 high ED foods/day (ED ≥3.0 kcal/g). Foods with an ED >1.0 kcal/g and <3.0 kcal/g will be unlimited; however, lowering the overall ED of the diet will be encouraged.
  Interventions: Behavioral: family-based obesity prevention lifestyle intervention
- STANDARD (Active Comparator): In the STANDARD condition participants will consume the recommendations for calories, fruits, vegetables and whole grains based on age and sex corresponding with MyPlate. The daily caloric recommendations from MyPlate are for weight maintenance.
  Interventions: Behavioral: family-based obesity prevention lifestyle intervention

INTERVENTIONS:
Behavioral: family-based obesity prevention lifestyle intervention — A family-based obesity prevention lifestyle intervention is based on the combination of behavioral therapy strategies, a physical activity prescription and a dietary prescription. Both the parent and child will be working to achieve the same behavioral targets.

SUMMARY:
This study investigates the effect of a low energy-density dietary prescription as compared to MyPlate recommendations in preschool children at risk for obesity.

ELIGIBILITY:
Inclusion Criteria:

* the parent is ≥18 years-old with a BMI ≥30 kg/m2 (indicating the child to be at risk for obesity);
* the child is 2-5 years-old with a BMI-for-age and sex <95th percentile;
* the parent and child live together ≥50% of the time;
* the parent and child are able to read, speak and understand English;
* the family has transportation to the University of Delaware; and
* the family is committed to the 6-month program.

Exclusion Criteria:

* the child is participating in a weight management program or seeing a Registered Dietitian for weight loss;
* the child is taking weight loss medication or medication that impacts appetite; or
* the child has a medical condition that impacts growth or has a medical condition that requires a specific eating plan.

Ages: 2 Years to 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 41 (Actual)
Dates: Start 2017-07-01 (Actual); Primary Completion 2021-11-09 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Dietary Energy Density | 6 months
  Dietary intake will be analyzed using NDSR and energy density (kcal/g) will be calculated.
Energy Intake | 6 months
  Dietary intake will be analyzed using NDSR and energy intake will be calculated.
Dietary Quality | 6 months
  Dietary intake will be analyzed using NDSR and used to calculate a Healthy Eating Index score.

SECONDARY OUTCOMES:
zBMI | 6 months
  A standardized z-score for BMI will be calculated based on the child's weight, height, age, and sex.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Delaware, Newark, Delaware, United States